CLINICAL TRIAL: NCT04151082
Title: Stop LCNP: High Dose Steroid Therapy for Late Radiation-Associated Lower Cranial Neuropathy: A Phase I/II Dose Finding Trial and Data Registry
Brief Title: High Dose Steroid Therapy (Prednisone or Methylprednisolone) for the Improvement of Symptoms of Late Radiation-Associated Lower Cranial Neuropathy in Oropharyngeal Cancer Survivors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0207; NCI-2019-06735 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0207 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-10-16; First posted 2019-11-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cranial Nerve Disorder; Head and Neck Carcinoma; Oropharyngeal Carcinoma
MeSH Terms: conditions — Cranial Nerve Diseases; Oropharyngeal Neoplasms | interventions — Methylprednisolone; exifone; Medrol Veriderm; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (steroid therapy) (Experimental): Patients receive prednisone PO (or by feeding tube) QD on days 1-5 and then taper off over 2 weeks or methylprednisolone IV over 1 hour on days 1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial studies the side effect and best dose of steroid therapy (prednisone or methylprednisolone) in improving symptoms of late radiation-associated lower cranial neuropathy in oropharyngeal cancer survivors. Steroid therapy with prednisone or methylprednisolone may help to improve symptoms associated with late radiation-associated lower cranial neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish feasibility and maximum tolerated dose (MTD) of steroid therapy that provides symptomatic improvement in oropharyngeal cancer (OPC) survivors with late lower cranial neuropathy (LCNP).

SECONDARY OBJECTIVE:

I. To examine endpoints that may be sensitive to functional or symptomatic gains with steroid therapy for late LCNP in OPC survivors by characterizing changes in symptoms, functional status, quality of life (QOL), neurophysiology, and imaging studies after steroid therapy.

TERTIARY OBJECTIVE:

I. To establish a hypothesis-generating database of physiologic, functional, and patient-reported outcomes (PROs) among head and neck cancer (HNC) survivors with late lower cranial neuropathy treated with steroid therapy.

OUTLINE: This is a phase I, dose-escalation study of steroid therapy followed by a phase II study.

Patients receive prednisone orally (PO) (or by feeding tube) once daily (QD) on days 1-5 and then taper off over 2 weeks or methylprednisolone intravenously (IV) over 1 hour on days 1-5 in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR CLINICAL TRIAL: Disease free adult survivors of oropharyngeal cancer
* INCLUSION CRITERIA FOR CLINICAL TRIAL: Treated with radiotherapy >= 2 years post treatment (disease status per surveillance imaging and clinical surveillance)
* INCLUSION CRITERIA FOR CLINICAL TRIAL: Late radiation-associated lower cranial neuropathy of XII with or without X nerve (LCNP cases will be considered therapy-related when imaging, physical examination, and/or biopsy fail to demonstrate structural or malignant source)
* INCLUSION CRITERIA FOR CLINICAL TRIAL: Willing and able to return for assessment post-steroid therapy
* INCLUSION CRITERIA FOR CLINICAL TRIAL: Able to complete symptom survey (MD Anderson Symptom Inventory - Head and Neck [MDASI-HN]) in validated languages: English, simplified Chinese, Filipino, Greek, Japanese, Korean, Russian, Spanish, Taiwanese
* INCLUSION CRITERIA FOR REGISTRY: Disease-free adult survivors of head and neck cancer
* INCLUSION CRITERIA FOR REGISTRY: >= 2 years post treatment (disease status per surveillance imaging and clinical surveillance)
* INCLUSION CRITERIA FOR REGISTRY: Late lower cranial neuropathy of XII with or without X nerve (LCNP cases will be considered therapy-related when imaging, physical examination, and/or biopsy fail to demonstrate structural or malignant source)
* INCLUSION CRITERIA FOR REGISTRY: Able to complete symptom survey (MDASI-HN) in validated languages: English, simplified Chinese, Filipino, Greek, Japanese, Korean, Russian, Spanish, Taiwanese

Exclusion Criteria:

* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Uncontrolled diabetes
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Uncontrolled hypertension (systolic > 160; diastolic > 90)
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Known gastrointestinal ulcer
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: History of psychosis
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Pregnant women
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Untreated or treatment refractory obstructive pharyngoesophageal stricture
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: Known history or diagnosis of bipolar disorder
* EXCLUSION CRITERIA FOR CLINICAL TRIAL: History of surgery near hypoglossal nerve path
* EXCLUSION CRITERIA FOR REGISTRY: Uncontrolled diabetes
* EXCLUSION CRITERIA FOR REGISTRY: Uncontrolled hypertension (systolic > 160; diastolic > 90)
* EXCLUSION CRITERIA FOR REGISTRY: Known gastrointestinal ulcer
* EXCLUSION CRITERIA FOR REGISTRY: History of psychosis
* EXCLUSION CRITERIA FOR REGISTRY: Pregnant women
* EXCLUSION CRITERIA FOR REGISTRY: Untreated or treatment refractory obstructive pharyngoesophageal stricture
* EXCLUSION CRITERIA FOR REGISTRY: Known history or diagnosis of bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 3 weeks
Change in MD Anderson Symptom Inventory - Head and Neck (MDASI-HN) top 5 mean | Baseline up to 3 weeks

SECONDARY OUTCOMES:
Improvement in tongue innervation on electromyography (EMG) findings | Up to 3 years
  1. EMG scores are based on a 4-point denervation potentials grade with '0' being 'none' and '4' being 'full interference patterns of potentials'.
  2. Nerve conduction study (NCS) scores are based on a 4-point scale ranging from 'none' (best) to 'severely prolonged' or 'severely reduced' (worst).
Improvement in dynamic imaging grade of swallowing toxicity (DIGEST) scores | Up to 3 years
  1. DIGEST scores are rated on a 0-4 scale from 0 (best) to 4 (worst).
Changes in maximum isometric lingual strength (MILS) and lingual range of motion (LROM) | Baseline up to 3 years
  1. MILS scores are rated on continuous scale from 0 (worst) to 100 (best).
  2. LROM scores are rated on an ordinal scale from 0 (worst) to 100 (best).
Changes in patient reported outcomes (PRO) on MD Anderson Dysphagia Inventory (MDADI), Performance Status Scale for Head and Neck (PSS-HN), or EuroQOL (EQ-5D) | Baseline up to 3 years
  1. MDADI scores are rated on a continuous scale from 20 (worst) to 100 (best).
  2. Diet, eating, and speech subscales of PSS-HN are rated on an ordinal scale from 0 (worst) to 100 (best).
  3. EQ-5D is rated on a continuous scale from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Hutcheson, BA,MS,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org